CLINICAL TRIAL: NCT05628376
Title: TRAcking Thoracic Cancer Evolution Through Therapy (Rx) EVO
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: UCL - 151927
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer, Non-small Cell; Small Cell Lung Cancer; Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, saliva, sputum, urine, stool, nasal curette
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: 300 participants with early stage resectable I-IIIB NSCLC
- Cohort B: 200 participants with unresectable late stage IIIB-IIIC or de novo metastatic (stage IV) NSCLC.
- Cohort C: 50-100 participants with stage I-IV SCLC or pleural mesothelioma.

SUMMARY:
TRACERx EVO is a programme of work using a prospective observational cohort study of participants with early- and late-stage non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC) and pleural mesothelioma.

DETAILED DESCRIPTION:
TRACERx EVO is a programme of work linked to an observational cohort study that consists of early and late-stage lung cancer and pleural mesothelioma. Participants will receive anti-cancer therapies (systemic therapies, radiotherapy and surgery, as per local and national guidelines). This study involves collecting a large amount of data, covering demographic and clinical characteristics, data throughout their follow up from the time of baseline/surgery, genomics and all other laboratory results using their blood, tissue, urine, saliva and stool samples. Data would also be retrieved from participant medical records. As such, there will be a wide range of analyses

ELIGIBILITY:
Inclusion Criteria:

* Cohort A, B and C :

  * Written Informed consent
  * Agreement to be followed up (including on-study assessments and sample collection) every 3 months in the first 2 years and then 6 monthly.
  * Agreement to be followed up at a TRACERx EVO site

Cohort A:

* Participants ≥18 years of age, with early stage I-IIIB NSCLC disease who are eligible for primary surgery
* Histopathologically confirmed NSCLC, or a strong suspicion of cancer on lung imaging necessitating surgery (e.g., diagnosis determined from frozen section in theatre)
* Primary surgery in keeping with NICE guidelines in (lobectomy, either open or thoracoscopic), lung parenchymal-sparing operations (segmentectomy or wedge resection) if a complete resection can be achieved, extensive surgery (bronchoangioplastic surgery, bilobectomy, pneumonectomy) if necessary to obtain clear margins, hilar and mediastinal lymph node sampling or en bloc resection)
* For participants proceeding with upfront primary surgery (i.e. no neoadjuvant therapy), a minimum tumour diameter at least 15mm to allow for sampling of at least two tumour regions
* Participants undergoing neoadjuvant treatment must have at least 1 region of fresh frozen or FFPE surgical or diagnostic biopsy tissue.
* Considered sufficiently fit for upfront standard of care primary surgery or neoadjuvant therapy if indicated
* Performance status 0 to 2

Cohort B:

* Participants ≥18 years of age, with late-stage unresectable stage IIIB and above NSCLC disease (TNM 8th edition) or presenting with stage IV de novo metastatic disease.
* Sufficient tissue (at least 1 region/biopsy), either FFPE or fresh frozen
* Deemed to be fit for anti-cancer treatment
* Performance status 0 to 2 Participants who were initially consented into Cohort A with a post-surgical staging of stage IIIB/C or IV could be included in Cohort B.

Cohort C:

* Participants ≥18 years of age, with any stage SCLC or pleural mesothelioma.
* Sufficient tissue (at least 1 region/biopsy), either FFPE or fresh frozen
* Deemed to be fit for anti-cancer treatment
* Performance status 0 to 2

Exclusion Criteria:

* Cohort A, B and C:

  * Other active malignancy
  * Any other* malignancy diagnosed or relapsed at any time, which is currently being treated (including by hormonal therapy).
  * Any other* current malignancy or malignancy diagnosed or relapsed within the past 3 years**.

    * *Exceptions are: non-melanomatous skin cancer, stage 0 melanoma in situ, and in situ cervical cancer
    * **An exception will be made for malignancies diagnosed or relapsed more than 2, but less than 3, years ago only if a pre-operative biopsy of the lung lesion has confirmed a diagnosis of NSCLC.
  * Psychological condition that would preclude informed consent
  * Diagnosis other than NSCLC, SCLC or pleural mesothelioma confirmed following surgery or biopsy
  * Confirmed diagnosis of known high-risk infections (e.g., Human Immunodeficiency Virus) (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection, tuberculosis and Creutzfeldt-Jacob disease) unless participant case is of a particular scientific interest and agreed in advance with research staff, local mortuary staff and pathologist.
  * Contra-indicated co-morbid conditions

Cohort A:

* Positive margins, incomplete resection or insufficient nodal sampling
* Insufficient tissue, i.e., for participants having upfront surgery and not having neoadjuvant therapy, a minimum of two tumour regions unlikely to be obtained for the study based on pre-operative imaging. For participants having neoadjuvant therapy i.e., at least one tissue biopsy to be obtained (Fresh Frozen or FFPE).
* Participant found to have pre-invasive lesions rather than invasive cancer following surgery, such as adenocarcinoma in situ or minimally invasive lesions will be withdrawn. However, the surgical tissue and baseline blood already collected will be sent to the central laboratory. These participants will not be followed-up in the study or required to provide any further blood samples. If these participants subsequently develop invasive cancer, the date of diagnosis and the tumour histology will be reported on the electronic data capture system.

Cohort B/C:

• Insufficient tissue, i.e., at least one tissue biopsy to be obtained (Fresh Frozen or FFPE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: I-IIIC or de novo metastatic (stage IV) Non-small cell lung cancer, stage I-IV Small cell lung cancer, pleural mesothelioma.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  DFS; recurrence or death from any cause): Cohorts A & C
Progression Free Survival | 5 years
  PFS; first disease progression or death from any cause): Cohorts B & C
Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No